CLINICAL TRIAL: NCT06952998
Title: Randomized Clinical Trial, Controlled With Conventional Treatment to Evaluate the Efficacy of Plasma Rich in Growth Factors (PRGF) in the Treatment of Foot Ulcers in Diabetic Patients With Peripheral Arterial Disease
Brief Title: Efficacy of Plasma Rich in Growth Factors (PRGF) in the Treatment of Foot Ulcers in Diabetic Patients With Peripheral Arterial Disease
Acronym: PIEDIABETICO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Biotechnology Institute IMASD (Industry)
Collaborators: Hospital de Basurto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTIIMD-01-EC-23-PIEDIABETICO
Record Dates: First submitted 2025-03-26; First posted 2025-05-01 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Foot Ulcers, Diabetic
MeSH Terms: conditions — Foot Ulcer | interventions — Intercellular Signaling Peptides and Proteins; Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical application of Plasma Rich in Growth Factors (PRGF) (Experimental): The Principal Investigator, or duly delegated qualified personnel, is responsible for the preparation using the KMU10-TPC Kit (BTI Biotechnology Institute, S.L.).
  Interventions: Drug: Topical application of Plasma Rich in Growth Factors (PRGF)
- Conventional treatment with adequate offloading and metabolic control, +/- antibiotic). (Active Comparator): Manufacturer: N/A
  Interventions: Procedure: Conventional treatment (conventional treatment with adequate offloading and metabolic control, +/- antibiotic).

INTERVENTIONS:
Drug: Topical application of Plasma Rich in Growth Factors (PRGF) — Topical application of PRGF will be maintained each time the patient undergoes the conventional treatment. The frequency of conventional treatment will be determined by the health specialist according to the evolution of the ulcer. The treatment will be maintained until complete wound closure or until the end of the follow-up period (6 months).
  Arms: Topical application of Plasma Rich in Growth Factors (PRGF)
Procedure: Conventional treatment (conventional treatment with adequate offloading and metabolic control, +/- antibiotic). — Conventional treatment (conventional treatment with adequate offloading and metabolic control, +/- antibiotic). The "TIME" dynamic wound closure strategy will be followed, which summarizes the four key points to stimulate the natural healing process: control of non-viable tissue, control of inflammation and infection, control of exudate and stimulation of the edges. After healing, chlorhexidine spray will be applied topically to these patients. The frequency of conventional treatment will be determined by the health specialist according to the evolution of the ulcer. Treatment will be maintained until complete wound closure or until the end of the follow-up period (6 months).
  Arms: Conventional treatment with adequate offloading and metabolic control, +/- antibiotic).

SUMMARY:
This study is a randomized clinical trial that compares the effectiveness of Plasma Rich in Growth Factors (PRGF) with conventional treatment for healing foot ulcers in diabetic patients who also have peripheral arterial disease. The goal is to assess how well PRGF promotes healing over a six-month period.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged at least 18 years
* Diagnosis of type 1 or 2 diabetes
* Presence of one or more ulcers below the malleoli
* Ulcer size ranging from 1 to 25 cm2
* Peripheral Arterial Disease (PAD)
* Meet at least 2 of the following crieria:
* Absence of peripheral pulses at any level on physical examination of lower extremities
* Ankle pressure of 50-90 mmHg
* Finger pressure 30-70 mmHg
* Ankle-branchial index (ABI) 0.5-0.9
* Finger-arm index (FIBI) 0.3-0.7
* Transcutaneous oxygen pressure (TcPO2) 30-59 mmHg
* Degree of infection of the lesion on IDSA/IWGDF scale not greater than 1
* Availability of observation during the study period
* Properly completed patient informed consent

Exclusion Criteria:

* Ulcers grade 3 or higher
* Positive markers for HCV, AfHBs, HIV-I/II or TP
* Diabetes mellitus with poor metabolic control (evidence of glycosylated hemoglobin >9%)
* Active systemic infection
* History of cancerous or precancerous lesions in the area of intervention
* On active treatment with other local treatment at the site of treatment
* On active treatment with immunosuppressants and/or other drugs contraindicating blood collection
* History of allergy to blood derivatives
* Previous diagnosis of coagulopathies
* Regular and continuous treatment (≥ 3 months) with NSAIDs (with the exception of the use of acetylsalicilic acid)
* Pregnancy or women of chilbearig age not taking effective contraceptive measures. These methods are, according to recommendations of the Clinical Trial Facilitation Group (CTFG) Contraception Working Group (CTFG) (V1.1), the following Hormonal contraception associated with ovulation inhibition, intrauterine decide (IUD), intrauterine hormone-releasing system, bilateral tubal ligation, vasectomy partner, sexual abstinence
* Breastfeeding women
* Treatment with monoclonal antibodies
* Any inabilities to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of ulcer healing evaluated with the RESVECH 2.0 index at six months | 6 months follow up
  RESVECH 2.0 (Expected Results of the Assessment and Evolution of Chronic Wound Healing Index). Composed of 6 variables whose psychometric properties are detailed as follows: reliability through internal consistency with a Cronbach's α of 0.63 and a Cronbach's α based on typed items of 0.72 (indicating greater consistency the closer α is to 1); with a content validity index for the total of the scale higher than 0.9, being called RESVECH2.0.
  These 6 final items that it assesses are:
  1. Injury dimensions
  2. Depth/tissues affected
  3. Edges
  4. Type of tissue in the wound bed
  5. Exudate
  6. Infection-inflammation (signs-biofilm) Thus, each of them receives a score, considering a total value of 0 for the healed ulcer, and reaching a maximum of 35 points as the worst possible wound as a result of the evaluation.

SECONDARY OUTCOMES:
Change in ulcer size at three and six months (percent) (area and depth) | 3 and 6 months follow up
  Change in ulcer size at three and six months (percent) (area and depth)
Frequency of ulcers with complete closure at three and six months (percent) | 3 and 6 months follow up
  Frequency of ulcers with complete closure at three and six months (percent)
Assessment of ulcer healing assessed with the RESVECH 2.0 index at baseline and at three months | Baseline and three months follow up
  RESVECH 2.0 (Expected Results of the Assessment and Evolution of Chronic Wound Healing Index). Composed of 6 variables whose psychometric properties are detailed as follows: reliability through internal consistency with a Cronbach's α of 0.63 and a Cronbach's α based on typed items of 0.72 (indicating greater consistency the closer α is to 1); with a content validity index for the total of the scale higher than 0.9, being called RESVECH2.0. These 6 final items that it assesses are: 1. Injury dimensions 2. Depth/tissues affected 3. Edges 4. Type of tissue in the wound bed 5. Exudate 6. Infection-inflammation (signs-biofilm) Thus, each of them receives a score, considering a total value of 0 for the healed ulcer, and reaching a maximum of 35 points as the worst possible wound as a result of the evaluation.
Assessment of amputation risk as measured by the WIfI scale at baseline, 3 and 6 months | Baseline, 3 and 6 months follow up
  The Wound, Ischemia, and foot Infection (WIfI) classification system assesses limb threat in three domains. Wound is graded 0-3 based on ulcer depth, extent, gangrene, and pain. Ischemia is graded 0-3 using ankle-brachial index, transcutaneous oxygen pressure, and toe pressure. Infection is graded 0-3 using adapted criteria from the IDSA and PEDIS systems. Each domain's score reflects severity, aiding in amputation risk and treatment planning.
Assessment of pain and quality of life at baseline, three and six months using the EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L) | Baseline, 3 and 6 months follow up
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS ranges from 0 (the worst health you can imagine) to 100 (the best health you can imagine), where higher scores represent better health outcomes
Evaluation of wound closure time | Throughout the study duration, assessed at each follow-up visit (up to 6 months post-enrollment)
  Evaluation of wound closure time
Safety endpoint. Incidence and type of adverse events | Throughout the study duration, assessed at each follow-up visit (up to 6 months post-enrollment)
  Incidence and type of adverse events
Safety endpoint. Presence of infetion at three and six months assessed with the IWGDF/IDSA classification | Throughout the study duration, assessed at each follow-up visit (up to 6 months post-enrollment)
  International Working Group on the Diabetic Foot (IWGDF) infectious diseases society of America (IDSA).
  Minimum Value: 1 (o "No Infection") Maximum Value: 4 (o "Severe Infection") Higher scores mean: Worse outcomes
Safety endpoint. Frequancy and type of deficiencies of the medical devices used for PRGF preparation. | Throughout the study duration, assessed at each follow-up visit (up to 6 months post-enrollment)
  Safety endpoint. Frequancy and type of deficiencies of the medical devices used for PRGF preparation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Basurto., Bilbao, Bizkaia, Spain